CLINICAL TRIAL: NCT05364866
Title: Cryoballoon Ablation Versus Medical Therapy in Patients With Atrial Fibrillation and Heart Failure With Different Ejection Fraction Categories
Brief Title: CAB Versus Medical Therapy in Patients With AF and HF With Different EF Categories
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-K039-01
Record Dates: First submitted 2022-04-06; First posted 2022-05-06 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical treatment group: Using class I or class III AAD to maintain sinus rhythm
  Interventions: Drug: Antiarrhythmic drug Therapy
- Cryoballoon ablation group: Pulmonary vein isolation by cryoballoon ablation using Medtronic Arctic Front Advance™ Cardiac CryoAblation Catheters (23mm and 28mm)
  Interventions: Device: cryoballoon ablation

INTERVENTIONS:
Drug: Antiarrhythmic drug Therapy — Propafenone, Sotalol and Amiodarone
  Other Names: Class I or III antiarrhythmic drug
  Groups: Medical treatment group
Device: cryoballoon ablation — Medtronic Arctic Front Advance™ Cardiac CryoAblation Catheters including 23mm and 28mm.
  Groups: Cryoballoon ablation group

SUMMARY:
This study is to assess the effectiveness and safety of cryoballoon ablation comparing with medical therapy in patients with atrial fibrillation and heart failure with different ejection fraction categories.

DETAILED DESCRIPTION:
Subjects with atrial fibrillation and heart failure with different ejection fraction categories are devided to either an anti-arrhythmic drug or cryoballoon catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with symptomatic paroxysmal or persistent atrial fibrillation：defined as at least two symptomatic episodes in the last six months prior to enrollment.
* At least 18 years old and not older than 80 years old.
* Able and willing to give informed consent.

Exclusion Criteria:

* History of AF treatment with class I or III AAD, including sotalol, with the intention to prevent an AF recurrence. However, patients pretreated with above AAD for less than 7 days with the intention to convert an AF episode are allowed.
* Previous left atrial ablation.
* Previous cardiac surgery including prosthetic valves.
* Permanent pacemaker or defibrillator implant.
* Second degree type II or third degree AV-block or a pattern of left/right bundle branch block.
* History of previous myocardial infarction or percutaneous intervention during the last 3 months.
* Any history of previous transient ischemic attack, prolonged reversible ischemic neurological deficit, and/or stroke.
* Known intracardiac thrombus formation.
* Pulmonary vein stent.
* Known cryoglobulinaemia.
* Active systemic infection.
* Hypertrophic cardiomyopathy.
* Life expectancy is ≤1 year.
* Reversible cause of atrial fibrillation (eg, hyperthyroidism or alcoholism).
* Abnormal long or short QT intervals, signs of Brugada syndrome, known family history of inherited ion channel disease, and/or arrhythmogenic right ventricular dysplasia.
* Chronic obstructive pulmonary disease with detected pulmonary hypertension and/or any other evidence of significant lung disease.
* Contraindication for oral anticoagulation.
* Pregnant women or woman of childbearing potential with inadequate birth control.
* Women who are breastfeeding.
* Any significant congenital heart defect corrected or not corrected; however, patent foramen ovale is allowed.
* Thrombocytosis (platelet count > 600,000/μL) or thrombocytopenia (platelet count < 100,000/μL).
* Untreated or uncontrolled hyperthyroidism or hypothyroidism.
* Renal dysfunction with glomerular filtration rate < 60 mL/min.
* Unstable angina pectoris.
* Symptomatic carotid stenosis.
* Myxoma based on laboratory abnormalities.
* Sarcoidosis.
* Unwilling to unable to comply with the study procedure and follow-up schedule due to any disease condition.
* Legal incapacity or evidence that the patient cannot understand the purpose and risks of the study, including inability to comply fully with study procedures and follow-up.
* Employed by Medtronic, or the department of an investigator, or close-familial relative of an investigator.
* Enrolled or planning to participate in a potentially confounding drug or device trial during this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with symptomatic paroxysmal or persistent atrial fibrillation：defined as at least two symptomatic episodes in the last six months prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment success at one year | one year
  Treatment success at 12 months after antiarrhythmic drug (AAD) initiation or ablation utilizing cryoballoon catheter measured by freedom from AF recurrence following a 3-month period after the index ablation or AAD initiation.
Rate of adverse events | one year
  Rate of complications and adverse events occurred during cryoballoon ablation and postoperative follow-up, including all-cause mortality, rehospitalisation for HF, and the composite event of all-cause mortality or HF hospitalisation

SECONDARY OUTCOMES:
Arrhythmia recurrence during blanking period | 3 months
  atrial tachycardia recurrence
Quality of life changes at 12 months measured by 12-Item Short Form Survey (SF-12) | one year
  The improvement in quality of life between baseline and 12 months after the index ablation procedure or AAD measured by 12-Item Short Form Survey (SF-12) with the values ranging from 12 - 47 (higher scores mean a worse outcome)
Quality of life changes at 12 months measured by AF Quality of Life Survey (AFEQT) | one year
  The improvement in quality of life between baseline and 12 months after the index ablation procedure or AAD measured by AF Quality of Life Survey (AFEQT) with the values ranging from 20 - 140 (higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT05364866/Prot_SAP_000.pdf